CLINICAL TRIAL: NCT06873230
Title: Assessment of Empathy Levels Among Dental Hygiene Students and Interns in Saudi Arabia: a Cross-Sectional Study
Brief Title: Assessment of Empathy Levels in Dental Hygiene Students and Interns
Acronym: Empathy
Status: Not yet recruiting | Type: Observational
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Dr Shiva Shankar Bugude, Assistant Professor, Qassim University
Other Study IDs: 421109786; capstone Project (Other: Qassim University, College of Applied Medical Sciences & Department of Public Health)
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Empathy
Keywords: Empathy; Dental Hygiene Students; Saudi Arabia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dental hygiene students and interns in Saudi Arabia: This research will employ a cross-sectional study design to assess empathy levels among dental hygiene students and interns in Saudi Arabia. The study will utilize the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS). Inclusion criteria:
  1. Dental hygiene students enrolled in accredited programs in Saudi Arabia.
  2. Dental hygiene interns currently working in dental clinics in Saudi Arabia.
  3. Dental hygiene students & interns who provide consent to participate in this online survey-based study.
  Exclusion criteria:
  1. Dental hygiene post-graduation student.
  2. Student who discontinued the program.
  3. Participants with any diagnosed neurological or psychiatric conditions that may significantly impact empathy (e.g., dementia, schizophrenia, autism spectrum disorder).
  4. Participants who have previously participated in similar research studies within the past 12 months.
  5. Dental hygiene students & interns who withdraw consent at any point during the study.
  Interventions: Other: The study will utilize the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) as the primary instrument for measuring empathy.

INTERVENTIONS:
Other: The study will utilize the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) as the primary instrument for measuring empathy. — This cross-sectional observational study utilizes the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) as the primary instrument for measuring empathy, distinguishing itself as the first of its kind to be conducted among Dental Hygiene students and interns in Saudi Arabia. The unique focus on this specific population in the Saudi context sets this research apart from previous studies in the field.

SUMMARY:
Empathy is a crucial element in the practice of dentistry, significantly influencing patient satisfaction and treatment outcomes. Recent studies have highlighted the importance of empathy in healthcare, suggesting that it is essential for effective clinician-patient communication and overall quality of care. Despite its recognized value, there is a concerning trend of declining empathy levels among dental students as they progress through their education. This decline may adversely affect their ability to connect with patients, ultimately impacting the quality of dental care provided.

In Saudi Arabia, research on empathy within dental education remains limited. A study conducted at King Abdulaziz University indicated that while dental students exhibited a sense of moral obligation, their overall empathy scores were lower than anticipated1. Furthermore, factors such as gender and academic year were found to influence empathy levels, with female students generally scoring higher than their male counterparts. Another study from Dammam reported similar findings, emphasizing the need for targeted interventions to enhance empathy among dental students and interns.

This proposed cross-sectional study aims to assess empathy levels among dental hygiene students and interns in Saudi Arabia. By utilizing the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS), this research will explore how demographic factors such as age, gender, and academic year correlate with empathy scores. The insights gained from this study could inform curriculum development and training programs aimed at fostering empathetic communication skills among future dental professionals.

DETAILED DESCRIPTION:
Research Hypothesis:

There is a significant difference in empathy levels among dental hygiene students and interns in Saudi Arabia, with factors such as gender, age, & academic year influencing empathy scores.

Null Hypothesis:

There is no significant difference in empathy levels among dental hygiene students and interns in Saudi Arabia, and factors such as gender, & academic year do not influence empathy scores.

Aims

1. To Quantitatively Measure Empathy Levels: Employ the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) to quantitatively assess the empathy levels of dental hygiene students and interns in Saudi Arabia.
2. To Investigate Demographic Correlates: Analyse the influence of demographic variables such as age, gender, academic year, and educational background on the empathy scores of dental hygiene students and interns.
3. To Compare Empathy Across Educational Stages: Examine differences in empathy levels between undergraduate dental hygiene students and those in internship positions to identify trends in empathetic development throughout their educational journey.
4. To Identify Factors Affecting Empathy: Explore how various factors, including prior academic performance and clinical exposure, may affect the empathy levels of dental hygiene students and interns.

Materials and methods:

Study design This research will employ a cross-sectional observational study design to assess empathy levels among dental hygiene students and interns in Saudi Arabia. The study will utilize the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) as the primary instrument for measuring empathy. Data will be collected at a single point in time, allowing for the evaluation of empathy scores in relation to various demographic factors. This design is appropriate for identifying the prevalence of empathy levels within the target population and exploring potential correlations with demographic variables. The study will adhere to ethical guidelines, ensuring informed consent is obtained from all participants prior to data collection.

Study setting:

The study will be conducted in various educational institutions across Saudi Arabia that offer dental hygiene programs. This includes both universities and colleges where dental hygiene students and interns are enrolled. The institutions will represent a diverse range of geographic locations and educational environments, ensuring a comprehensive assessment of empathy levels among the target population. Data collection will take place during the academic year, allowing for the inclusion of students from different academic stages, including first-year students and those in internship positions.

Sample size or Population of interest:

The population of interest for this study comprises dental hygiene students and interns enrolled in accredited dental hygiene programs across Saudi Arabia. Due to the lack of specific enrolment data for dental hygiene students in 2024, sample size determination was based on previous studies examining empathy levels in healthcare education within the country.

Based on existing literature, a sample size of approximately 200 participants is deemed sufficient to achieve statistical power for detecting significant differences in empathy scores. This estimate is informed by similar studies conducted in Saudi Arabia, which have successfully utilized comparable sample sizes to assess empathy among healthcare students. For instance, a study by Naguib et al. (2022) assessed empathy levels among dental interns and postgraduate students with a sample size of 250 participants9. Another study by Alhassan et al. (2021) evaluated empathy among dental students with a sample size of 30010. These references support the feasibility of recruiting a similar number of participants for the current study.

Sampling technique:

This study will employ a snowball sampling technique, a non-probability sampling method, to recruit participants among dental hygiene students and interns in Saudi Arabia. This non-probability sampling method is selected for its efficacy in reaching populations that are difficult to access through conventional random sampling methods. Initially, a small group of participants will be identified through direct outreach to dental hygiene programs at selected institutions. These participants will then be asked to refer their peers, thereby facilitating the recruitment of additional subjects within the target population.

To mitigate potential biases associated with snowball sampling, several strategies will be implemented:

1. Initiate multiple "seed" points across different geographical areas to enhance sample diversity.
2. Diverse Initial Contacts: The initial participants will be selected from various academic years and institutions to ensure a diverse representation of the population. This approach aims to minimize homogeneity in the sample and enhance the generalizability of the findings.
3. Inclusion Criteria: Clear inclusion criteria will be established to ensure that only current dental hygiene students and interns are recruited. This will help maintain the relevance of the sample to the research objectives.
4. Monitoring Referrals: The referral process will be monitored to avoid clustering of responses from similar individuals or groups. Participants will be encouraged to refer individuals from different backgrounds and experiences.
5. Anonymity and Confidentiality: Assuring participants of their anonymity and confidentiality may encourage more honest responses, thereby reducing bias related to social desirability.

By implementing these strategies, the study aims to enhance the validity of the findings while effectively utilizing the snowball sampling method to reach a broader population of interest.

Data collection procedure:

Data for this study will be collected through an online survey administered via Google Forms, utilizing the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS) as the primary instrument for measuring empathy levels among dental hygiene students and interns.

1. Introduction and Consent: The survey will begin with an introduction outlining the purpose of the study, emphasizing the importance of empathy in dental hygiene practice and patient care. Participants will be informed that their responses will remain confidential and anonymous. Following this, a consent form will be presented, requiring participants to confirm their willingness to participate in the study before proceeding.
2. Demographic and Academic Information: The survey will include sections to collect demographic information such as age, gender, academic year, and educational institution. This data will help contextualize the empathy scores and identify any correlations with demographic variables.
3. Jefferson Scale of Empathy (JSE-HPS): The core component of the survey will consist of the JSE-HPS questionnaire, which includes 20 items designed to assess various dimensions of empathy in health profession students. Participants will respond to each item using a 7-point Likert scale, ranging from "strongly agree" to "strongly disagree." This self-report format allows participants to reflect on their empathetic attitudes and behaviors in clinical settings.

The collected data will be analyzed quantitatively to determine empathy levels among participants and explore potential associations with demographic factors.

Data Collection Steps:

1. Questionnaire Pilot Testing: The survey questionnaire will be available in both Arabic and English and will undergo a pilot test with 20 dental hygiene students and 20 dental hygiene interns to assess clarity and validity prior to distribution.
2. Initial Recruitment of Seed Participants: The first "seed" participants will be recruited through dental hygiene departments at universities, professional dental organizations in Saudi Arabia, and relevant online professional networks.
3. Distribution of the Questionnaire: Seed participants will receive an anonymized link to the Google Form, accompanied by an introductory message that outlines the study's objectives, procedures, and ethical considerations, including anonymity, confidentiality, and voluntary participation.
4. Snowball Sampling: Seed participants will be encouraged to share the link with other eligible dental hygienists within their networks, promoting further dissemination through email, messaging applications, and social media platforms.
5. Data Collection Timeline: Data collection will take place over a specified period (e.g., 4-6 weeks), with periodic reminder messages sent to participants.
6. Data Management Procedures: Responses collected via Google Forms will be automatically stored in a secure Google Sheet. After anonymization-removing direct identifiers and assigning study IDs-the data will be exported for analysis.

Pilot study:

To enhance the quality and effectiveness of our main research study, we conducted a pilot survey involving 20 dental hygiene students & 20 dental hygiene interns.

Data management and analysis plan.

In view of Data protection & Data management following measures will be taken:

1. Anonymization and De-identification
2. Secure Data Storage by possible encryption
3. Data Access Control
4. Data Backup and Recovery
5. Documentation and Record Keeping

Data will be analyzed by biostatistician using statistical software SPSS. The variables in the study and will be checked for their associations using appropriate tests of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Dental hygiene students enrolled in accredited programs in Saudi Arabia.
2. Dental hygiene interns currently working in dental clinics in Saudi Arabia.
3. Dental hygiene students & interns who provide consent to participate in this online survey-based study.

Exclusion Criteria:

1. Dental hygiene post-graduation student.
2. Student who discontinued the program.
3. Participants with any diagnosed neurological or psychiatric conditions that may significantly impact empathy (e.g., dementia, schizophrenia, autism spectrum disorder).
4. Participants who have previously participated in similar research studies within the past 12 months.
5. Dental hygiene students & interns who withdraw consent at any point during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of interest for this study comprises dental hygiene students and interns enrolled in dental hygiene programs across Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Overall Empathy Score | The observational study will involve data collection from participants between March and May 2025, with a total study duration of two months.
  The main outcome is the quantitative measure of empathy using the Jefferson Scale of Empathy-Health Profession Students (JSE-HPS). This involves:
  Total Score: A composite score derived from all 20 items on the JSE-HPS, which reflects the overall empathy level of each participant.

SECONDARY OUTCOMES:
Demographic Correlations | The observational study will involve data collection from participants between March and May 2025, with a total study duration of two months.
  Analysis of how empathy scores vary with key demographic variables collected in the study:
  Age: Comparing empathy levels across different age groups. Gender: Evaluating differences between male and female participants. Academic Stage: Assessing variations in empathy between undergraduate dental hygiene students and interns. This comparison may highlight trends in empathy development as students progress in their clinical training.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banu AM, Ursoniu S, Gotia SL, Putnoky S, Serban CL. Understanding empathy and theory of mind in Romanian dental students for improved educational strategies. Sci Rep. 2025 Jan 31;15(1):3880. doi: 10.1038/s41598-025-88264-1. PMID 39890985
- [Background] Collins DM, Iannucci JM, Townsend JA, Kearney RC. Predictors of Empathy Among Dental Hygiene Undergraduate Students. J Dent Hyg. 2024 Aug;98(4):20-27. PMID 39137992
- [Background] Detsomboonrat P, Theppanich S, Banyen S, Hongviphat S, Khamnil Y, Lapauthaya K, Somboonsavatdee A, Min SN. Empathy level towards patients among thai dental students: a cross-sectional study. BMC Oral Health. 2023 Mar 30;23(1):184. doi: 10.1186/s12903-023-02891-6. PMID 36997938